CLINICAL TRIAL: NCT00122850
Title: A Comparison of Duloxetine Hydrochloride, Venlafaxine Extended Release, and Placebo in the Treatment of Generalized Anxiety Disorder.
Brief Title: A Comparison of Duloxetine Hydrochloride, Marketed Comparator, and Placebo in the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 7107; F1J-MC-HMDU
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride; Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine
Drug: venlafaxine
Drug: placebo

SUMMARY:
This study will examine duloxetine compared with placebo and an active comparator in the treatment of generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients at least 18 years of age, presenting with generalized anxiety disorder (GAD) based on the disease diagnostic criteria. Must suffer from GAD and not from an adjustment disorder or anxiety disorder not otherwise specified. The symptoms of GAD should not be situational in nature.

Exclusion Criteria:

* Any current and primary DSM-IV Axis I diagnosis other than GAD, including:

  * Patients diagnosed with major depressive disorder within the past 6 months; or
  * Patients diagnosed with panic disorder, or post-traumatic stress disorder within the past year; or
  * Patients diagnosed with obsessive-compulsive disorder, bipolar affective disorder, psychosis, factitious disorder, or somatoform disorders during their lifetimes.
* The presence of an Axis II disorder or history of antisocial behavior, which, in the judgement of the investigator, would interfere with compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2004-10; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To assess whether duloxetine hydrochloride 60 to 120 mg once daily is superior to placebo in the treatment of GAD during a 10-week, double-blind acute therapy phase, defined as statistically greater reduction in anxiety symptoms as measured by the HAMA.

SECONDARY OUTCOMES:
Self-reported anxiety symptomatology;Quality of Life;Clinical Global Improvement;HAMA factor scores

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oakbrook Terrace, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Florence, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cambridge, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seattle, Washington

REFERENCES:
- [Derived] Perlis RH, Fijal B, Dharia S, Houston JP. Pharmacogenetic investigation of response to duloxetine treatment in generalized anxiety disorder. Pharmacogenomics J. 2013 Jun;13(3):280-5. doi: 10.1038/tpj.2011.62. Epub 2012 Jan 17. PMID 22249355
- [Derived] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Derived] Allgulander C, Nutt D, Detke M, Erickson J, Spann M, Walker D, Ball S, Russell J. A non-inferiority comparison of duloxetine and venlafaxine in the treatment of adult patients with generalized anxiety disorder. J Psychopharmacol. 2008 Jun;22(4):417-25. doi: 10.1177/0269881108091588. PMID 18635722
- [Derived] Allgulander C, Hartford J, Russell J, Ball S, Erickson J, Raskin J, Rynn M. Pharmacotherapy of generalized anxiety disorder: results of duloxetine treatment from a pooled analysis of three clinical trials. Curr Med Res Opin. 2007 Jun;23(6):1245-52. doi: 10.1185/030079907X182202. Epub 2007 Apr 25. PMID 17559726
- [Derived] Endicott J, Russell JM, Raskin J, Detke MJ, Erickson J, Ball SG, Marciniak M, Swindle RW. Duloxetine treatment for role functioning improvement in generalized anxiety disorder: three independent studies. J Clin Psychiatry. 2007 Apr;68(4):518-24. doi: 10.4088/jcp.v68n0405. PMID 17474806
- [Derived] Hartford J, Kornstein S, Liebowitz M, Pigott T, Russell J, Detke M, Walker D, Ball S, Dunayevich E, Dinkel J, Erickson J. Duloxetine as an SNRI treatment for generalized anxiety disorder: results from a placebo and active-controlled trial. Int Clin Psychopharmacol. 2007 May;22(3):167-74. doi: 10.1097/YIC.0b013e32807fb1b2. PMID 17414743
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com